CLINICAL TRIAL: NCT04089462
Title: Effects of Frequency and Duration of Exercise in People With Type 1 Diabetes - A Randomized Crossover Study
Brief Title: Effects of Frequency and Duration of Exercise in People With Type 1 Diabetes A Randomized Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-19035830
Record Dates: First submitted 2019-09-05; First posted 2019-09-13 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 1; Insulin Hypoglycemia
Keywords: Exercise; Insulin pump; Diabetes Mellitus, Type 1; Guidelines
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Intervention Model Description: An open-labelled randomized controlled crossover study will be performed. The participants will go through the following elements:
  1. Screening day
  2. Run-in period
  3. Intervention period
  4. Wash-out period
  5. Intervention period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. "Five sessions per period" - "Two sessions per period" (Other)
  Interventions: Behavioral: "Five sessions per period" - "Two sessions per period"
- 2. "Two sessions per period" - "Five sessions per period" (Other)
  Interventions: Behavioral: "Two sessions per period" - "Five sessions per period"

INTERVENTIONS:
Behavioral: "Five sessions per period" - "Two sessions per period" — Period 1: 5 exercise sessions on 5 consecutive days (4 min anaerobic exercise and 30 min aerobic exercise per session)
  Period 2: 2 exercise sessions within a 5-day period (10 min anaerobic exercise and 75 min aerobic exercise per session)
  Arms: 1. "Five sessions per period" - "Two sessions per period"
Behavioral: "Two sessions per period" - "Five sessions per period" — Period 1: 2 exercise sessions within a 5-day period (10 min anaerobic exercise and 75 min aerobic exercise per session)
  Period 2: 5 exercise sessions on 5 consecutive days (4 min anaerobic exercise and 30 min aerobic exercise per session)
  Arms: 2. "Two sessions per period" - "Five sessions per period"

SUMMARY:
According to the Standards of Medical Care in Diabetes by the American Diabetes Association, people with diabetes should aim for 30 minutes of moderate-to-vigorous intensity aerobic exercise at least 5 days a week or a total of 150 minutes per week and doing some type of strength training at least 2 times per week in addition to aerobic activity. However, the effects of different forms and intervals of exercise on glycemic control are not well established. Exercise increases the risk of hypoglycemia both during and several hours after exercise.

There are several strategies to avoid hypoglycemia during exercise. The most common strategy is to reduce insulin and to take carbohydrates before the exercise starts. Short-acting insulin analogs have a duration of approximately four hours, thus reductions need to be planned and done well in advance before the exercise starts. Since different types of exercise (aerobic, strength training or high intensity training) affect blood glucose in different ways and most exercise sessions include a combination of the types, these strategies are often associated with difficulties in obtaining stable blood glucose. The American Diabetes Association guidelines do not explicitly recommend a daily workout routine but outline recommendations for weekly amounts of exercise as there is currently insufficient evidence on the ideal timing, frequency and duration of exercise for preventing hypoglycemia.

Hypothesis: in people with type 1 diabetes, time in hypoglycemia can be reduced if exercise is performed daily over five consecutive days compared to the same total amount of exercise performed at 2 days with at least 2 days interval.

Aim: to evaluate the impact of the same total amount of exercise split into either five consecutive sessions or two sessions with at least 2 days in between on percentage of time spent in hypoglycemia and other glycemic parameters in people with type 1 diabetes.

DETAILED DESCRIPTION:
The participants will go through two interventions: Exercise one session per day for five consecutive days and Exercise one session per day for two days within five days. The exercise session will start with anaerobic (push-ups, back-curls, sit-ups, triceps-dips and jumps) exercise followed by aerobic exercise (moderate intensity of running, walking or cycling). Between the two intervention periods, there will be a wash-out period.

Intervention: 'Exercise one session per day for five consecutive days'. Duration per session: Anaerobic: 4 min, Aerobic: 30 min. Sessions per intervention period: Five. Total duration per intervention period: Anaerobic: 20 min. Aerobic: 150 min. Total: 170 min

Intervention:Exercise one session per day for two days within five days. Duration per session: Anaerobe: 10 min, Aerobe: 75 min. Sessions per intervention period: 2. Total duration per intervention period: Anaerob: 20 min Aerobe: 150 min Total: 170 min

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes ≥ 2 year
* Insulin pump ≥ 1 year.
* Use of carbohydrate counting and the insulin pump bolus calculator for all meals

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), per oral or injected corticosteroids or other drugs affecting glucose metabolism during the intervention period or within 30 days prior to study start
* Known or suspected alcohol or drug abuse
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the participant unsuitable for study participation
* Females who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Inability to understand the participants' information and to give informed consent
* Chronic use or unable to stop acetaminophen (paracetamol) use
* Allergy to the patch of CGM
* Hypoglycemia unawareness, quantified by Pedersen-Bjergaard
* Severe hypoglycemia within the last year
* Vigorous-intensity exercise for more than 60 minutes on 3 days or more per week

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the hypoglycemic range (CGM <3.9 mmol/l) | The primary intervention period from 06:00h study day 1 - 06:00h study day 6 (ITT)
  Intention-to-treat analysis (ITT).

SECONDARY OUTCOMES:
Percentage of time spent in the hypoglycemic range (CGM <3.9 mmol/l) | Primary intervention period from 06:00h study day 1 - 06:00h study day 6 PP
  Per protocol analysis (PP)
Percentage of time spent in the alert and clinical hypoglycemic range | Study day 1: The day when the first exercise session is performed and registered.
  Level 1 (alert): CGM or SMBG value of 3.0-3.9 mmol/l with or without symptoms. Level 2 (clinical): CGM or SMBG value of < 3.0 mmol/l with or without symptoms. Outcome is compared between the two intervention periods in a per protocol analysis (PP) and intention-to-treat analysis (ITT)
Percentage of time spent in the alert and clinical hypoglycemic range | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Level 1 (alert): CGM or SMBG value of 3.0-3.9 mmol/l with or without symptoms. Level 2 (clinical): CGM or SMBG value of < 3.0 mmol/l with or without symptoms. Outcome is also compared between the two intervention periods in a per protocol analysis (PP) and intention-to-treat analysis (ITT)
Percentage of time spent in the alert and clinical hypoglycemic range | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Level 1 (alert): CGM or SMBG value of 3.0-3.9 mmol/l with or without symptoms. Level 2 (clinical): CGM or SMBG value of < 3.0 mmol/l with or without symptoms. Outcome is also compared between the two intervention periods in a per protocol analysis (PP) and intention-to-treat analysis (ITT)
Percentage of time spent in the alert and clinical hypoglycemic range | Day time: 06:00-22:00h from during study day 1 to study day 6.
  Level 1 (alert): CGM or SMBG value of 3.0-3.9 mmol/l with or without symptoms. Level 2 (clinical): CGM or SMBG value of < 3.0 mmol/l with or without symptoms. Outcome is also compared between the two intervention periods in a per protocol analysis (PP) and intention-to-treat analysis (ITT)
Percentage of time spent in the alert and clinical hypoglycemic range | Night time: 22:00-06:00h from during study day 1 to study day 6.
  Level 1 (alert): CGM or SMBG value of 3.0-3.9 mmol/l with or without symptoms. Level 2 (clinical): CGM or SMBG value of < 3.0 mmol/l with or without symptoms. Outcome is compared between the two intervention periods in a per protocol analysis (PP) and intention-to-treat analysis (ITT)
Percentage of time spent in the alert and clinical hypoglycemic range | The time the participant has recorded start and end of exercise session during study day 1 to study day 6
  Level 1 (alert): CGM or SMBG value of 3.0-3.9 mmol/l with or without symptoms. Level 2 (clinical): CGM or SMBG value of < 3.0 mmol/l with or without symptoms. Outcome is compared between the two intervention periods in a per protocol analysis (PP) and intention-to-treat analysis (ITT)
Number of alert and clinical hypoglycemia events | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Number of alert and clinical hypoglycemia events | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Number of alert and clinical hypoglycemia events | Day time: 06:00-22:00h during study day 1 - study day 6
  Per protocol analysis and intention-to-treat analysis
Number of alert and clinical hypoglycemia events | Night time: 22:00-06:00h during study day 1 - study day 6
  Per protocol analysis and intention-to-treat analysis
Number of alert and clinical hypoglycemia events | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 study day 6
  Per protocol analysis and intention-to-treat analysis
Number of severe hypoglycemia events during | Study day 1: The day when the first exercise session is performed and registered
  Per protocol analysis and intention-to-treat analysis
Number of severe hypoglycemia events | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Number of severe hypoglycemia events | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Number of severe hypoglycemia events | Day time: 06:00-22:00h during study day 1 - study day 6
  Per protocol analysis and intention-to-treat analysis
Number of severe hypoglycemia events | Night time: 22:00-06:00h during study day 1 - study day 6
  Per protocol analysis and intention-to-treat analysis
Number of severe hypoglycemia events | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 - study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in range (3.9-10 mmol/l) | Study day 1: The day when the first exercise session is performed and registered
  Per protocol analysis and intention-to-treat analysis
Percentage of time in range (3.9-10 mmol/l) | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Percentage of time in range (3.9-10 mmol/l) | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Percentage of time in range (3.9-10 mmol/l) | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in range (3.9-10 mmol/l) | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in range (3.9-10 mmol/l) | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in good range (3.9-7.8 mmol/l) | Study day 1: The day when the first exercise session is performed and registered.
  Per protocol analysis and intention-to-treat analysis
Percentage of time in good range (3.9-7.8 mmol/l) | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Percentage of time in good range (3.9-7.8 mmol/l) | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Percentage of time in good range (3.9-7.8 mmol/l) | Day time: 06:00-22:00h and Night time: 22:00-06:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in good range (3.9-7.8 mmol/l) | Exercise time: The time the participant has recorded start and end of exercise session during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in hyperglycemia (>10 mmol/l) | Study day 1: The day when the first exercise session is performed and registered.
  Per protocol analysis and intention-to-treat analysis
Percentage of time in hyperglycemia (>10 mmol/l) | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Percentage of time in hyperglycemia (>10 mmol/l) | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in hyperglycemia (>10 mmol/l) | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in hyperglycemia (>10 mmol/l) | Exercise time: The time the participant has recorded start and end of exercise session during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Percentage of time in hyperglycemia (>10 mmol/l) during all the predefined time blocks. Per protocol analysis and intention-to-treat analysis | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Glycemic variability measured as standard deviation (SD), coefficient of variation (CV) and low and high blood glucose index (LBGI/HBGI) during all the predefined time blocks in the intervention period | Study day 1: The day when the first exercise session is performed and registered.
  Per protocol analysis and intention-to-treat analysis
Glycemic variability measured as standard deviation (SD), coefficient of variation (CV) and low and high blood glucose index (LBGI/HBGI) during all the predefined time blocks in the intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Glycemic variability measured as standard deviation (SD), coefficient of variation (CV) and low and high blood glucose index (LBGI/HBGI) during all the predefined time blocks in the intervention period | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Glycemic variability measured as standard deviation (SD), coefficient of variation (CV) and low and high blood glucose index (LBGI/HBGI) during all the predefined time blocks in the intervention period | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Glycemic variability measured as standard deviation (SD), coefficient of variation (CV) and low and high blood glucose index (LBGI/HBGI) during all the predefined time blocks in the intervention period | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Mean CGM glucose level du during all the predefined time blocks in the intervention period | Study day 1: The day when the first exercise session is performed and registered.
  Per protocol analysis and intention-to-treat analysis
Mean CGM glucose level du during all the predefined time blocks in the intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Mean CGM glucose level du during all the predefined time blocks in the intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Mean CGM glucose level du during all the predefined time blocks in the intervention period | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Mean CGM glucose level du during all the predefined time blocks in the intervention period | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Mean CGM glucose level du during all the predefined time blocks in the intervention period | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
CGM estimated eA1c during the primary intervention period | The Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Total carbohydrate intake registered from the insulin pumps during all the predefined time blocks in the intervention period | Study day 1: The day when the first exercise session is performed and registered.
  Per protocol analysis and intention-to-treat analysis
Total carbohydrate intake registered from the insulin pumps during all the predefined time blocks in the intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Total carbohydrate intake registered from the insulin pumps during all the predefined time blocks in the intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Total carbohydrate intake registered from the insulin pumps during all the predefined time blocks in the intervention period | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Total carbohydrate intake registered from the insulin pumps during all the predefined time blocks in the intervention period | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Total carbohydrate intake registered from the insulin pumps during all the predefined time blocks in the intervention period | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Carbohydrate interventions for prevention and treatment of hypoglycemia registered by the participants in the booklet for the primary and total intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis c) Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
Carbohydrate interventions for prevention and treatment of hypoglycemia registered by the participants in the booklet for the primary and total intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis c) Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
Change in total daily insulin dose (basal and bolus insulin) of 7 days prior to screening day and during the primary and total intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Change in total daily insulin dose (basal and bolus insulin) of 7 days prior to screening day and during the primary and total intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Actigraph wrist wear time during all predefined time blocks | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Actigraph wrist wear time during all predefined time blocks | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Actigraph wrist wear time during all predefined time blocks | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Actigraph wrist wear time during all predefined time blocks | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Actigraph wrist wear time during all predefined time blocks | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Physical activity energy expenditure (accelerometer and heart rate based) measured as kcal during all predefined time blocks | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Physical activity energy expenditure (accelerometer and heart rate based) measured as kcal during all predefined time blocks | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Physical activity energy expenditure (accelerometer and heart rate based) measured as kcal during all predefined time blocks | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Physical activity energy expenditure (accelerometer and heart rate based) measured as kcal during all predefined time blocks | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Physical activity energy expenditure (accelerometer and heart rate based) measured as kcal during all predefined time blocks | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Metabolic expenditure rate for the primary intervention periods | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Metabolic expenditure rate for the primary intervention periods | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Number of exercise (light to vigorous) and sedentary bouts in the primary intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Number of exercise (light to vigorous) and sedentary bouts in the primary intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time in sedentary during predefined time blocks | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time in sedentary during predefined time blocks | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Time in sedentary during predefined time blocks | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Time in sedentary during predefined time blocks | Night time: 22:00-06:00h during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Time in sedentary during predefined time blocks | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Time in light physical activity during predefined time blocks | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time in light physical activity during predefined time blocks | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Time in light physical activity during predefined time blocks | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Time in light physical activity during predefined time blocks | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Time in moderate physical activity during predefined time blocks | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time in moderate physical activity during predefined time blocks | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days).
  Per protocol analysis and intention-to-treat analysis
Time in moderate physical activity during predefined time blocks | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Time in moderate physical activity during predefined time blocks | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Time in vigorous physical activity during predefined time blocks | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time in vigorous physical activity during predefined time blocks | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time in vigorous physical activity during predefined time blocks | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Time in vigorous physical activity during predefined time blocks | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Number of steps during predefined time blocks | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Number of steps during predefined time blocks | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Number of steps during predefined time blocks | Day time: 06:00-22:00h during study day 1-study day 6
  Per protocol analysis and intention-to-treat analysis
Number of steps during predefined time blocks | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Heart rate during exercise sessions | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
R-R intervals during exercise sessions (f) | Exercise time: The time the participant has recorded start and end of exercise session during study day 1 -study day 6
  Per protocol analysis and intention-to-treat analysis
Sleep latency (min) during the primary and total intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Sleep latency (min) during the primary and total intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Total sleep time (min) during the primary and total intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Total sleep time (min) during the primary and total intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Sleep efficiency (%) during the primary and total intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Sleep efficiency (%) during the primary and total intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Number of awakening during sleep in the primary and total intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Number of awakening during sleep in the primary and total intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time of awakening during sleep in the primary and total intervention period | Primary intervention period: 06:00h study day 1 - 06:00h study day 6 (= 5 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Time of awakening during sleep in the primary and total intervention period | Secondary intervention period: 08:00h day 1 - 08:00h day 8 (= 7 x 24-hour days)
  Per protocol analysis and intention-to-treat analysis
Question about patient preference regarding the two study arms | At the end of study. Study day 6 the last interventions period.
  Per protocol analysis and intention-to-treat analysis

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle IK Steineck, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data are processed and merged into at least one scientific article published in international peer-reviewed scientific journal. Positive, negative and inconclusive results will be published as soon as scientifically justifiable.
Supporting Information: Study Protocol, SAP
Time Frame: 21 oktober 2020

REFERENCES:
- [Derived] Steineck IIK, Ranjan AG, Schmidt S, Norgaard K. Time spent in hypoglycemia is comparable when the same amount of exercise is performed 5 or 2 days weekly: a randomized crossover study in people with type 1 diabetes. BMJ Open Diabetes Res Care. 2021 Jan;9(1):e001919. doi: 10.1136/bmjdrc-2020-001919. PMID 33509935